CLINICAL TRIAL: NCT00006929
Title: A Phase I/II Study of Carboplatin / Paclitaxel / Suramin Chemotherapy in Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Suramin, Paclitaxel, and Carboplatin in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01403; OSU 0045; OSU-0045; OSU-00HO224; NCI-2250; CDR0000068345; U01CA076576 (NIH)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Suramin; Carboplatin; Paclitaxel; Taxes

ARMS (1):
- Treatment (suramin, paclitaxel, carboplatin) (Experimental): Patients receive suramin IV over 30 minutes on days 1 and 2. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: suramin; Drug: carboplatin; Drug: paclitaxel; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: suramin — Given IV
  Other Names: 309 F; Antrypol; Bayer 205; Fourneau 309; Germanin
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining suramin, paclitaxel, and carboplatin in treating patients who have stage IIIB or stage IV non-small cell lung cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the minimum effective dose of suramin that will reduce resistance to chemotherapy with paclitaxel and carboplatin in patients with stage IIIB or IV non-small cell lung cancer (phase I). (Phase I closed to accrual 1/29/02).

II. Evaluate pharmacokinetic interactions of this drug combination in these patients (phase I). (Phase I closed to accrual 1/29/02).

III. Determine the objective response rate in patients treated with this regimen (phase II [chemotherapy-naive patients closed to accrual 9/1/03]).

IV. Determine the time to tumor progression, progression-free rate at 6 months, and 1-year survival of patients treated with this regimen (phase II [chemotherapy-naive patients closed to accrual 9/1/03]).

OUTLINE: Patients in phase II are stratified according to prior treatment (chemotherapy naive [closed to accrual 9/1/03] vs chemotherapy refractory). Phase I (phase I closed to accrual 1/29/02):

Patients receive suramin IV over 30 minutes on days 1 and 2. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of suramin until the target dose is determined. The target dose is defined as the dose at which at least 5 of 6 patients achieve optimal plasma concentrations of suramin and no more than 1 of 6 patients exceed optimal level. Doses of paclitaxel are adjusted until the maximum tolerated dose in combination with suramin and paclitaxel is determined.

Phase II (chemotherapy-naive patients closed to accrual 9/1/03): Patients receive the target dose of suramin IV over 30 minutes on days 1 and 2. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3-6 weeks.

PROJECTED ACCRUAL: Approximately 82 patients (18 for phase I [phase I closed to accrual 1/29/02] and 64 for phase II [chemotherapy-naive patients closed to accrual 9/1/03]) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced non-small cell lung cancer

  * Stage IIIB not amenable to concurrent chemotherapy or radiotherapy (e.g., pleural effusion or low pulmonary reserve)
  * Stage IV
* Measurable disease
* Meets criteria for 1 of the following:

  * Chemotherapy naive (phases I and II) (phase I closed to accrual 1/29/02) (phase II [chemotherapy-naive patients] closed to accrual 9/1/03)
  * Previously treated (phase I) (phase I closed to accrual 1/29/02)

    * Received no more than 1 prior chemotherapy regimen
  * Chemotherapy refractory, defined as disease progression during or within 3 months after carboplatin/paclitaxel chemotherapy (phase II)
* No known brain or leptomeningeal disease unless previously irradiated, currently not undergoing corticosteroid therapy, and clinically asymptomatic
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 9.0 g/dL
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 50 mL/min
* Calcium less than 11.5 mg/dL
* No history of myocardial infarction within the past 6 months
* No history of congestive heart failure requiring therapy
* No history of unstable angina
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active serious infection
* HIV negative
* No concurrent uncontrolled diabetes mellitus
* No known hypersensitivity to Cremophor EL
* No grade 2 or greater neuropathy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No known psychiatric condition that would preclude study compliance
* At least 28 days since prior cytotoxic chemotherapy and recovered
* Prior radiotherapy allowed except to indicator lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2000-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of suramin of 10-20 uM (Phase I) | Up to 72 hours
Objective response rate (complete response [CR] and partial response [PR]) according to Response Evaluation Criteria in Solid Tumors (RECIST) (Phase II) | Up to 4 years

SECONDARY OUTCOMES:
Progression-free survival according to RECIST (Phase II) | At 6 months
Survival (Phase II) | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villalona-Calero, Principal Investigator — Ohio State University
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States